CLINICAL TRIAL: NCT06975111
Title: Focusing on the Menopausal Transition to Improve Mid-Life Women's Health
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-0943; U1111-1322-1036 (Other: World Health Organization)
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Menopause; Menopause Hot Flashes; Menopause Related Conditions; Cardiovascular
MeSH Terms: interventions — Metformin; semaglutide; Antihypertensive Agents; Angiotensin Receptor Antagonists; fezolinetant

STUDY DESIGN:
Intervention Model Description: Participants will be placed into treatment interventions based on their health and screening tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Preventative Health Advice (Experimental): Participants will be given preventative health advice and asked to wear an activity & sleep monitor.
  Interventions: Behavioral: Life style intervention; Drug: Fezolinetant; Drug: Hormonal therapy
- At Risk for Heart Disease (Active Comparator): Medications will be given to each participant in this arm that lowers your heart disease risk.
  Interventions: Drug: Metformin; Drug: Anti-hypertensives; Drug: Lipid Lowering Medication; Behavioral: Life style intervention
- Overweight Women (Active Comparator): Women who fit in this category will receive medication for lowering insulin resistance and/or a weight loss medication.
  Interventions: Drug: Metformin; Drug: semaglutide
- Women with Obesity (Active Comparator): Women that are over a BMI of 30 kg/m2 will be offered a GLP-1 antagonist.
  Interventions: Drug: semaglutide
- Women With Hot Flashes (Active Comparator): Women with Hot flashes will have either hormonal or non-hormonal medication to reduce the number and/or severity of hot flashes.
  Interventions: Drug: Fezolinetant; Drug: Hormonal therapy

INTERVENTIONS:
Drug: Metformin — Metformin will be given to participants who have a elevated HbA1c and also for weightloss.
  Arms: At Risk for Heart Disease; Overweight Women
Drug: semaglutide — Overweight women and women with obesity will take Semaglutide for weight-loss
  Arms: Overweight Women; Women with Obesity
Drug: Anti-hypertensives — a. Antihypertensives, with the goal of maintaining blood pressure at 130/80 or lower per ACC guidelines19. Per current clinical guidelines and standard of care, hypertension will be treated first with monotherapy using either an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB), a calcium channel blocker, or a thiazide diuretic provided that are no contraindications.
  Other Names: The use of angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB), a calcium channel blocker, or a thiazide diuretic.
  Arms: At Risk for Heart Disease
Drug: Lipid Lowering Medication — . First line agents will be generic statin medications (atorvastatin or rosuvastatin)whichever is covered by the participant's health insurance), barring contraindication to their use.
  Other Names: The use of generic statins
  Arms: At Risk for Heart Disease
Behavioral: Life style intervention — will simply be followed and given preventive advice (maintenance of a normal BMI and physical activity, moderation in salt intake, and no more than 1 alcoholic drink per day). They will be provided with a wearable activity monitor. This advice will be based on guidelines by the American Heart Association and the Menopause Society.
  Arms: At Risk for Heart Disease; Preventative Health Advice
Drug: Fezolinetant — Women with menopausal symptoms will be treated with hormone therapy (estrogen and progesterone) if appropriate, or with a neurokinin receptor antagonist (Fezolinetant). This can be treatment for women in any arm of the study as well as an arm by its self.
  Arms: Preventative Health Advice; Women With Hot Flashes
Drug: Hormonal therapy — Participants will be treated with estrogen and/or progesterone for treatment of hot flashes in women during the study.
  Arms: Preventative Health Advice; Women With Hot Flashes

SUMMARY:
What if midlife women, who are inherently at an increased risk for future cardiometabolic disease due to transitioning into menopause, had access to a suite of evidence-based health interventions? Could these interventions reduce menopause-related inflammation, restore a healthier cardiometabolic profile, reverse epigenetic aging, and reduce bothersome menopausal symptoms? The ultimate goal of this work is to attenuate future disease and enhance women's quality of life, extend healthspan and increase productivity.

ELIGIBILITY:
Inclusion Criteria:

* aged 45-55
* In the late menopausal transition, defined as 60 days of amenorrhea but less than 365 days of amenorrhea18
* No current use of hormone therapy or hormonal contraception
* Presence of a uterus and at least one ovary in order to track menstrual patterns
* Have a smartphone and broadband access adequate to accept telehealth appointments

Exclusion Criteria:

* Lack of broadband access (activity and survey data will be collected electronically whenever possible and some visits will be via telehealth)
* Lack of regular menstrual periods in mid-reproductive life (ages 25-38) when not on hormones or not pregnant.
* Pregnancy or actively trying to get pregnant
* Inability to adhere to study protocol schedule
* Untreated alcoholism
* Un- Diagnosed abnormal uterine bleeding
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia (MEN 2) for participants with a BMI> 30 kg/m2.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are studying the menopausal transition which only happens in women.
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic aging measurements of "PhenoAge" | Up to 2 years
  Change in epigenetic aging, as assessed by PhenoAge. PhenoAge calculates a biological age score based on key biomarkers circulating in the bloodstream. A lower PhenoAge score suggests slower biological aging, while a higher score indicates accelerated aging.
Epigenetic aging measurements of "GrimAge" | Up to 2 years
  Epigenetic aging, as assessed by GrimAge. GrimAge assesses lifespan from examining DNA Methylation.

SECONDARY OUTCOMES:
IL-1 | Up to 2 years
  Inflammatory IL-1 serum levels, examined to determine a person's inflammatory state. Higher levels of IL-1 can indicate more inflammation. Being in an "inflamed state" can have detrimental effects on a woman's health.
TNF-alpha | Up to 2 years
  Serum inflammatory marker TNF-alpha. Higher levels of TNF-alpha can indicate more inflammation. TNF-alpha is examined to determine a person's inflammatory state.
IL-6 | Up to 2 years
  Serum IL-6 levels. IL-6 is examined to determine a person's inflammatory state. Higher levels of IL-6 indicate more inflammation. Being in an "inflamed state" can have detrimental effects on a women's health.
IL-8 | Up to 2 years
  IL-8 serum levels. IL-8 is examined to determine a person's inflammatory state. Higher levelf of IL-8 indicate more inflammation. Being in an "inflamed state" can have detrimental effects on a women's health.
Flow-mediated dilation | Up to 2 years
  Flow-mediated dilation measures the diameter of vascular and endothelial cell function and predicts cardiovascular event risk. The diameter of the target artery is measured by high-resolution external vascular ultrasound in response to an increase in blood flow.
Serum Marker for Ovarian Aging | Up to 2 years
  Anti-mullerian hormones (AMH) serum levels will be analyzed. AMH is an indicator of ovarian aging and reflects egg supply. Lower levels of AMH indicate a lower egg supply.
MENQOL survey | Up to 2 years
  Menopause-specific Quality of Life (MENQOL) measures quality of life in menopausal women. It is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor, psychosocial, physical, and sexual. There will be a overall score and we are examining if there is a change in response to treatment.
Eaotoxin levels | Up to 2 years
  Eaotoxin is a inflammatory marker that increases when there is an inflammed state in a woman. Serum Eaotoxin will be measured before, during and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado-School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will share the information but have not developed the exact plan to share. All information and data will be de-identified prior to sharing. To share the data we will require a proposal detailing the use if IPD.

REFERENCES:
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Greendale GA, Huang MH, Wight RG, Seeman T, Luetters C, Avis NE, Johnston J, Karlamangla AS. Effects of the menopause transition and hormone use on cognitive performance in midlife women. Neurology. 2009 May 26;72(21):1850-7. doi: 10.1212/WNL.0b013e3181a71193. PMID 19470968
- [Background] Matthews KA, Crawford SL, Chae CU, Everson-Rose SA, Sowers MF, Sternfeld B, Sutton-Tyrrell K. Are changes in cardiovascular disease risk factors in midlife women due to chronological aging or to the menopausal transition? J Am Coll Cardiol. 2009 Dec 15;54(25):2366-73. doi: 10.1016/j.jacc.2009.10.009. PMID 20082925
- [Background] Samargandy S, Matthews KA, Brooks MM, Barinas-Mitchell E, Magnani JW, Janssen I, Kazlauskaite R, El Khoudary SR. Abdominal visceral adipose tissue over the menopause transition and carotid atherosclerosis: the SWAN heart study. Menopause. 2021 Mar 1;28(6):626-633. doi: 10.1097/GME.0000000000001755. PMID 33651741
- [Background] Tanaka T, Basisty N, Fantoni G, Candia J, Moore AZ, Biancotto A, Schilling B, Bandinelli S, Ferrucci L. Plasma proteomic biomarker signature of age predicts health and life span. Elife. 2020 Nov 19;9:e61073. doi: 10.7554/eLife.61073. PMID 33210602
- [Background] Thurston RC, Carroll JE, Levine M, Chang Y, Crandall C, Manson JE, Pal L, Hou L, Shadyab AH, Horvath S. Vasomotor Symptoms and Accelerated Epigenetic Aging in the Women's Health Initiative (WHI). J Clin Endocrinol Metab. 2020 Apr 1;105(4):1221-7. doi: 10.1210/clinem/dgaa081. PMID 32080740
- [Background] Fahy GM, Brooke RT, Watson JP, Good Z, Vasanawala SS, Maecker H, Leipold MD, Lin DTS, Kobor MS, Horvath S. Reversal of epigenetic aging and immunosenescent trends in humans. Aging Cell. 2019 Dec;18(6):e13028. doi: 10.1111/acel.13028. Epub 2019 Sep 8. PMID 31496122
- [Background] Thurston RC, Aslanidou Vlachos HE, Derby CA, Jackson EA, Brooks MM, Matthews KA, Harlow S, Joffe H, El Khoudary SR. Menopausal Vasomotor Symptoms and Risk of Incident Cardiovascular Disease Events in SWAN. J Am Heart Assoc. 2021 Feb 2;10(3):e017416. doi: 10.1161/JAHA.120.017416. Epub 2021 Jan 20. PMID 33470142
- [Background] Hedderson MM, Liu EF, Lee C, El Khoudary SR, Gold EB, Derby CA, Thurston RC. Vasomotor Symptom Trajectories and Risk of Incident Diabetes. JAMA Netw Open. 2024 Oct 1;7(10):e2443546. doi: 10.1001/jamanetworkopen.2024.43546. PMID 39480425
- [Background] Cho L, Davis M, Elgendy I, Epps K, Lindley KJ, Mehta PK, Michos ED, Minissian M, Pepine C, Vaccarino V, Volgman AS; ACC CVD Womens Committee Members. Summary of Updated Recommendations for Primary Prevention of Cardiovascular Disease in Women: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 May 26;75(20):2602-2618. doi: 10.1016/j.jacc.2020.03.060. PMID 32439010
- [Background] Patel D, Ayesha IE, Monson NR, Klair N, Patel U, Saxena A, Hamid P. The Effectiveness of Metformin in Diabetes Prevention: A Systematic Review and Meta-Analysis. Cureus. 2023 Sep 28;15(9):e46108. doi: 10.7759/cureus.46108. eCollection 2023 Sep. PMID 37900422
- [Background] Santoro N, Kuhn K, Pretzel S, Schauer IE, Fought A, D'Alessandro A, Stephenson D, Bradford AP. A high-fat eucaloric diet induces reprometabolic syndrome of obesity in normal weight women. PNAS Nexus. 2023 Dec 18;3(1):pgad440. doi: 10.1093/pnasnexus/pgad440. eCollection 2024 Jan. PMID 38178979
- [Background] Legro RS, Hansen KR, Diamond MP, Steiner AZ, Coutifaris C, Cedars MI, Hoeger KM, Usadi R, Johnstone EB, Haisenleder DJ, Wild RA, Barnhart KT, Mersereau J, Trussell JC, Krawetz SA, Kris-Etherton PM, Sarwer DB, Santoro N, Eisenberg E, Huang H, Zhang H; Reproductive Medicine Network. Effects of preconception lifestyle intervention in infertile women with obesity: The FIT-PLESE randomized controlled trial. PLoS Med. 2022 Jan 18;19(1):e1003883. doi: 10.1371/journal.pmed.1003883. eCollection 2022 Jan. PMID 35041662
- [Background] Tannous A, Bradford AP, Kuhn K, Fought A, Schauer I, Santoro N. A randomised trial examining inflammatory signaling in acutely induced hyperinsulinemia and hyperlipidemia in normal weight women-the reprometabolic syndrome. PLoS One. 2021 Mar 25;16(3):e0247638. doi: 10.1371/journal.pone.0247638. eCollection 2021. PMID 33764994
- [Background] Mogul HR, Freeman R, Nguyen K, Frey M, Klein LA, Jozak S, Tanenbaum K. Carbohydrate modified diet & insulin sensitizers reduce body weight & modulate metabolic syndrome measures in EMPOWIR (enhance the metabolic profile of women with insulin resistance): a randomized trial of normoglycemic women with midlife weight gain. PLoS One. 2014 Sep 26;9(9):e108264. doi: 10.1371/journal.pone.0108264. eCollection 2014. PMID 25259787
- [Background] Mogul H, Freeman R, Nguyen K. METFORMIN-SUSTAINED WEIGHT LOSS AND REDUCED ANDROID FAT TISSUE AT 12 MONTHS IN EMPOWIR (ENHANCE THE METABOLIC PROFILE OF WOMEN WITH INSULIN RESISTANCE): A DOUBLE BLIND, PLACEBO-CONTROLLED, RANDOMIZED TRIAL OF NORMOGLYCEMIC WOMEN WITH MIDLIFE WEIGHT GAIN. Endocr Pract. 2016 May;22(5):575-86. doi: 10.4158/EP151087.OR. Epub 2016 Jan 20. PMID 26789348
- [Background] "The 2022 Hormone Therapy Position Statement of The North American Menopause Society" Advisory Panel. The 2022 hormone therapy position statement of The North American Menopause Society. Menopause. 2022 Jul 1;29(7):767-794. doi: 10.1097/GME.0000000000002028. PMID 35797481
- [Background] Simpson DJ, Chandra T. Epigenetic age prediction. Aging Cell. 2021 Sep;20(9):e13452. doi: 10.1111/acel.13452. Epub 2021 Aug 20. PMID 34415665
- [Background] Karlamangla AS, Shieh A, Greendale GA. Hormones and bone loss across the menopause transition. Vitam Horm. 2021;115:401-417. doi: 10.1016/bs.vh.2020.12.016. Epub 2021 Jan 29. PMID 33706956
- [Background] Moreau KL, Hildreth KL, Klawitter J, Blatchford P, Kohrt WM. Decline in endothelial function across the menopause transition in healthy women is related to decreased estradiol and increased oxidative stress. Geroscience. 2020 Dec;42(6):1699-1714. doi: 10.1007/s11357-020-00236-7. Epub 2020 Aug 8. PMID 32770384
- [Background] Janssen I, Powell LH, Crawford S, Lasley B, Sutton-Tyrrell K. Menopause and the metabolic syndrome: the Study of Women's Health Across the Nation. Arch Intern Med. 2008 Jul 28;168(14):1568-75. doi: 10.1001/archinte.168.14.1568. PMID 18663170
- [Background] El Khoudary SR, Wildman RP, Matthews K, Thurston RC, Bromberger JT, Sutton-Tyrrell K. Progression rates of carotid intima-media thickness and adventitial diameter during the menopausal transition. Menopause. 2013 Jan;20(1):8-14. doi: 10.1097/gme.0b013e3182611787. PMID 22990755
- [Background] Bromberger JT, Epperson CN. Depression During and After the Perimenopause: Impact of Hormones, Genetics, and Environmental Determinants of Disease. Obstet Gynecol Clin North Am. 2018 Dec;45(4):663-678. doi: 10.1016/j.ogc.2018.07.007. Epub 2018 Oct 25. PMID 30401549
- [Background] El Khoudary SR, Greendale G, Crawford SL, Avis NE, Brooks MM, Thurston RC, Karvonen-Gutierrez C, Waetjen LE, Matthews K. The menopause transition and women's health at midlife: a progress report from the Study of Women's Health Across the Nation (SWAN). Menopause. 2019 Oct;26(10):1213-1227. doi: 10.1097/GME.0000000000001424. PMID 31568098